CLINICAL TRIAL: NCT03229070
Title: Cycle-ergometer in the Postoperative of Thoracic Surgery: A Randomized, Controlled Clinical Trial Comparing the Effect of Interval Training With Continuous Training on Performance in the Six-minute Walk Test
Brief Title: Cycle-ergometer in the Postoperative of Thoracic Surgery
Acronym: CE_PTS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Collaborators: Irmandade Santa Casa de Misericórdia de Porto Alegre (Other)
Responsible Party: Principal Investigator, Fabrício Edler Macagnan, PhD, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cycle-ergometer- PTS 2017
Record Dates: First submitted 2017-07-21; First posted 2017-07-25 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Functional Capacity; Fatigue; Dyspnea; Muscle Strength
Keywords: Thoracic Surgery; Postoperative Period; Rehabilitation; Early mobilization; Cycle-ergometer
MeSH Terms: conditions — Fatigue; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): Control Group: Pre-surgical evaluations (Six-minute walk test, sit and lift test 30 in seconds, and Piper fatigue scale) and assessments at discharge
- Interval effort group (Experimental): Interval effort group: Pre-surgical evaluations (Six-minute walk test, sit and lift test 30 in seconds, and Piper fatigue scale) Active phase (high load) lasting 60 seconds, followed by an active recovery phase with light / moderate load (60% of the maximum load) lasting 4 minutes. The pedaling speed should be maintained between 30-60rpm. There will be 5 cycles that will total 20 minutes of physical effort, and assessments at discharge.
  Interventions: Other: Interval effort group
- Continuous effort group (Experimental): Pre-surgical evaluations (Six-minute walk test, sit and lift test 30 in seconds, and Piper fatigue scale) Intensity used will be mild / moderate, ie 60% of the maximum load reached in the incremental test. The pedaling speed should be maintained between 30-60rpm. The execution time, from this exercise regime will be 20 minutes, and assessments at discharge.
  Interventions: Other: Continuous effort group

INTERVENTIONS:
Other: Interval effort group — Pre-surgical evaluations (Six-minute walk test, sit and lift test 30 in seconds, and Piper fatigue scale) Active phase (high load) lasting 60 seconds, followed by an active recovery phase with light / moderate load (60% of the maximum load) lasting 4 minutes. The pedaling speed should be maintained between 30-60rpm. There will be 5 cycles that will total 20 minutes of physical effort, and assessments at discharge.
  Arms: Interval effort group
Other: Continuous effort group — Pre-surgical evaluations (Six-minute walk test, sit and lift test 30 in seconds, and Piper fatigue scale) Intensity used will be mild / moderate, ie 60% of the maximum load reached in the incremental test. The pedaling speed should be maintained between 30-60rpm. The execution time, from this exercise regime will be 20 minutes, and assessments at discharge.
  Arms: Continuous effort group

SUMMARY:
Post-lateral thoracotomies and assisted thoracic surgery (CTVA) are the main surgical approaches for pulmonary resections. One of the counterpoints of these surgical approaches is postoperative pain, which in addition to causing ventilatory changes and reduction of lung capacities, contributes to bed rest and consequent decrease in patients' functionality. These complications increase hospitalization time and hospital costs, being determinant factors for perioperative morbidity and mortality. In order to prevent these outcomes of reduce the functional capacity of patients, new physiotherapeutic approaches have been adopted, such as the use of the cycloergometer. Recent studies show that the early use of this device brings benefits such as: improved blood circulation and venous return, increased muscle strength, improved functional capacity and reduced symptoms of dyspnea and fatigue. This study aims to compare the effect of interval training with continuous cycle ergometer training on performance in the six-minute walk test. Randomized and controlled clinical trial performed with patients submitted to elective thoracic surgery, hospitalized at the intensive care unit (ICU) and in the hospitalization unit of the Hospital Pavilhão Pereira Filho of the Santa Casa de Misericórdia Brotherhood of Porto Alegre. Participants will be randomized into three groups: control group (CG), interval exercise group (GHG) and continuous exercise group (GEC). Functional capacity assessments will be performed through the six-minute walk test (6MWT) and the chair sit and lift (TSL) test in 30 seconds, and evaluation of the clinical state of fatigue through the revised Piper-Fatigue Scale. The evaluations will be performed preoperatively and at hospital discharge.

DETAILED DESCRIPTION:
Will include patients between 30 and 80 years of age, of both sexes, submitted to thoracic surgery with incision by posterolateral thoracotomy, as well as those submitted to video-assisted thoracic surgery for pulmonary resection (bulectomy, segmentectomy, lobectomy, pneumectomy).

The cycloergometer rehabilitation program will be performed twice a day for 20 minutes.

The expectation of comparing two different types of muscle overload (interval training versus continuous training) is that the training of shorter duration and greater load also has a greater demand on the cardiopulmonary system of these patients and, therefore, a better response to the functional capacity rehabilitation program of these individuals.

ELIGIBILITY:
Inclusion Criteria:

* Patients submitted to thoracic surgery with postero-lateral thoracotomy incision, as well as those submitted to video-assisted thoracic surgery for pulmonary resection (bulectomy, segmentectomy, lobectomy, pneumectomy);
* Subjects extubated;
* Hemodynamically stable (mean arterial pressure (MAP) between 60 mmHg and 100 mmHg, heart rate (HR) between 50 bpm and 110 bpm
* Peripheral oxygen saturation ≥ 90%;
* With prescription for respiratory and motor physiotherapy.

Exclusion Criteria:

* Individuals who are not extubated for up to 6 hours in the immediate postoperative period, who require a second procedure during the immediate postoperative period;
* Alterations in cognitive function;
* Severe and decompensated cardiac arrhythmias;
* Hypotensive crisis;
* Hemoptysis;
* Chest bleeding requiring reintervention;
* sepsis;
* Need for reintubation;
* Signs of ventilatory effort;
* Acute renal failure;
* Unstable angina or malignant arrhythmias;
* Fever.
* Fluid drainage greater than 300 ml in the first six hours
* Or those who refuse to participate in the study.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2017-08-26 (Estimated); Primary Completion 2017-12-30 (Estimated); Study Completion 2018-02-28 (Estimated)

PRIMARY OUTCOMES:
Maximum distance performed on six-minute test | 6 minutes
  Walk in a 30m corridor

SECONDARY OUTCOMES:
Maximum number of times you succeed lift and sit on the chair | 30 seconds
  With your arms crossed against your chest, sit up and get up from the chair

IPD SHARING:
Plan to Share IPD: No